CLINICAL TRIAL: NCT02975960
Title: Adipose Tissue-derived Mesenchymal Stem Cells for Cell-based Therapy in the Treatment of Systemic Sclerosis
Brief Title: ADMSCs for the Treatment of Systemic Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Collaborators: Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Jung Hee Koh, Clinical Professor, Principal Investigator, The Catholic University of Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KC16TISI0343
Record Dates: First submitted 2016-11-09; First posted 2016-11-29 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Systemic Sclerosis
Keywords: systemic sclerosis; adipose derived stem cell; stromal vascular fraction; digital ulcer; gangrene
MeSH Terms: conditions — Scleroderma, Systemic; digital ulcers; Gangrene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stromal vascular fraction injection (Experimental): Injection of autologous stromal vascular fraction on hand.
  Interventions: Biological: injection of autologous stromal vascular fraction

INTERVENTIONS:
Biological: injection of autologous stromal vascular fraction — 1. Acquiring autologous stromal vascular fraction (SVF) from liposuction
  2. purifying SVF from lipoaspirates and making syringe filled with SVF
  3. SVF injection - Inject SVF on fingers subcutaneously.

SUMMARY:
Systemic sclerosis (SSc) is a rare autoimmune disease, mainly characterized by cutaneous and visceral fibrosis. Digital ulcer and sclerosing skin are commonly affected on hands, but the treatment for these manifestations are often ineffective.

Adipose tissue contains stromal vascular fraction (SVF), which is abundant multipotent stem cells, capable of tissue repair. A prior study (NCT01813279) has shown the safety and tolerance at 6 months of the subcutaneous injection of SVF in the fingers in SSc.

There are only few ways to manage SSc patients with skin lesion who already have treated with several medications (including vasodilators, PDE5 inhibitor, endothelin receptor antagonist) but some times their skin lesions are critical physically and emotionally.

Autologous SVF injection could be one of the treatment options to treat skin lesion of SSc. Thus, the investigators study the efficacy and potential adverse event in Korean patients with SSc.

DETAILED DESCRIPTION:
In this study, the investigators will inject autologous Stromal vascular fraction.

1) Acquiring autologous stromal vascular fraction by plastic surgeon

1. Liposuction
2. Extraction and purifying SVF using Smart-X system (15-20 min)
3. Making syringe filled with autologous SVF

2) SVF injection

Inject SVF subcutaneously with 25G needle in finger

ELIGIBILITY:
Inclusion Criteria:

1. Patients who fulfill 2013 American college of Rheumatology/ European League Against Rheumatism Criteria for the classification of systemic sclerosis.
2. The skin lesion was not improved after 6 months treatment with conventional therapy.

Exclusion Criteria:

1. Pregnancy
2. Start new medications within 3 months prior to enrollment
3. Previous sympathectomy or amputation
4. Current systemic infection
5. AIDS, Syphilis, hepatitis B&C
6. BMI <17kg/m2
7. Cognitive dysfunction and other psychologic problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-10-25 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2018-01-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline modified Rodnan Skin score (mRSS) of hands at 12 weeks | baseline, 12 weeks
  Assess hands mRSS

SECONDARY OUTCOMES:
Change from baseline Raynaud's condition score at 12 weeks | baseline, 12 weeks
  The severity (frequency and intensity of crises) of Raynaud's phenomenon
Change from baseline Visual Analog Score for pain the hands at 12 weeks | baseline, 12 weeks
  Patient report hand pain degree, comparing baseline and 12 weeks
Changes from baseline mRSS (total) at 12 weeks | baseline, 12 weeks
  Assess total mRSS (including hands)
Change from baseline Kapandji score at 12weeks | baseline, 12 weeks
  assess the mobility of both hands
Change from baseline Cochin hand function scale at 12 weeks | baseline, 12 weeks
  Assess hand function (patients reported outcome)
Change from baseline Systemic sclerosis HAQ at 12 weeks | baseline, 12 weeks
  he quality of life- score adapted to systemic sclerosis
Change from baseline peripheral vasculature at 12 weeks | baseline, 12 weeks
  Assess peripheral vascularity by Nailfold capillaroscopy
Change from baseline finger circumference at 12 weeks | baseline, 12 weeks
  Measure second to fifth finger circumference

CONTACTS AND LOCATIONS:
Overall Officials: Jung Hee Koh, MD, Principal Investigator — Seoul St.Mary's hospital, The Catholic university of Korea
Locations (1):
- Seoul St. Mary's hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No